CLINICAL TRIAL: NCT03174236
Title: First Line Antimicrobials in Children With Complicated Severe Acute Malnutrition
Acronym: FLACSAM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: University College, London (Other); London School of Hygiene and Tropical Medicine (Other); Swansea Trials Unit (Unknown); Kenya Medical Research Institute (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEMRI/SERU/CGMR-C/063/3399; 1-17 (Other: OxTREC); 105431/Z/14/Z (Other Grant/Funding Number: Joint Global Health Trials, MRC/DfID/Wellcome Trust)
Record Dates: First submitted 2017-05-15; First posted 2017-06-02 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Malnutrition Severe; Antibiotic Resistance; Antibiotic Toxicity
MeSH Terms: interventions — Ceftriaxone; Penicillin G; Metronidazole; Gentamicins

STUDY DESIGN:
Intervention Model Description: The trial will investigate two separate antimicrobial interventions in a 2x2 factorial design randomised controlled clinical trial. A factorial design allows more than one intervention to be tested and is useful in assessing a potential package of care. Two randomisations will be made. The two interventions will be analysed separately. Ceftriaxone and metronidazole is an effective and commonly used antibiotic combination, hence major interactions that interfere with efficacy are considered unlikely. However, evidence for interaction between the two interventions will be tested.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Metronidazole and its placebo will be masked. They will both be contained in similar bottles labelled with sequential study numbers according to a prepared blocked randomisation list before the trial begins. They will also be of similar appearance.
  Ceftriaxone and penicillin + gentamicin will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ceftriaxone (Experimental): Arm 1 IV Ceftriaxone: Participants in this group receive 80mg/kg IV ceftriaxone once a day for a minimum of 48 hours and a usual maximum of seven days.
  Interventions: Drug: Ceftriaxone
- Benzyl penicillin plus gentamicin (Active Comparator): Arm 2 IV Benzyl penicillin plus gentamicin (usual care): Participants in this group receive 50 000 U/kg IV benzyl penicillin every six hours for a minimum of two days and a maximum of seven days.
  Interventions: Drug: Benzyl penicillin; Drug: Gentamicin
- Metronidazole (Experimental): Arm 1 Metronidazole: Participants receive 10 to 16 mg/kg oral metronidazole twice a day for seven days.
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Arm 2 Placebo: Participants receive an oral placebo dose to match that for Metronidazole twice a day for seven days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ceftriaxone — Ceftriaxone a third-generation cephalosporin. Ceftriaxone is active against a broad spectrum of Gram positive and Gram negative bacteria.
  Arms: Ceftriaxone
Drug: Benzyl penicillin — The currently recommended first-line antibiotics for the treatment of severe acute malnutrition are gentamicin plus ampicillin or penicillin.
  Arms: Benzyl penicillin plus gentamicin
Drug: Metronidazole — The WHO guidelines recommend that Metronidazole may be given in addition to broad-spectrum antibiotics, "however, the efficacy of this treatment has not been established in clinical trials."
  Arms: Metronidazole
Other: Placebo — Suspension manufactured to match metronidazole
  Arms: Placebo
Drug: Gentamicin — The currently recommended first-line antibiotics for the treatment of severe acute malnutrition are gentamicin plus ampicillin or penicillin.
  Arms: Benzyl penicillin plus gentamicin

SUMMARY:
Children with severe malnutrition who are admitted sick to hospitals have a high mortality(death rate), usually because of infection. All children with severe malnutrition admitted to hospitals are treated with antibiotics(medication used to kill bacteria). However, the current antibiotics used in hospitals may not be the most effective. It is possible that the antibiotics that are currently used after initial antibiotics should be used first. No studies have been carried out to determine if the current antibiotics used for treating malnourished children who are sick and admitted in hospital are the most appropriate. The aim of this study is to find out if a changed antibiotic system for children with malnutrition is safe, reduces the risk of death and improves nutritional recovery.

DETAILED DESCRIPTION:
Children with complicated severe acute malnutrition (SAM) admitted to hospital in sub-Saharan Africa have a case fatality(death rate) between 12% and more than 20%. Because children with SAM may not exhibit the usual signs of infection, WHO guidelines recommend routine antibiotics(medication used to kill bacteria). However, this is based on "low quality evidence". There is evidence that because of bacterial resistance to the currently recommended first-line antibiotics (gentamicin plus ampicillin or penicillin) could be less effective than potential alternatives. Some hospitals in Africa are already increasing use of ceftriaxone as a first-line treatment. However, this is not based on any data that ceftriaxone actually improves outcomes. Of concern is that ceftriaxone use may also lead to increased antimicrobial resistance, including inducing extended spectrum beta-lactamase (ESBL) and other classes of resistance.

A further area where evidence for policy is lacking is the use of metronidazole in severely malnourished children. The WHO guidelines recommend "Metronidazole 7.5 mg/kg every 8 h for 7 days may be given in addition to broad-spectrum antibiotics; however, the efficacy of this treatment has not been established in clinical trials." Metronidazole is effective against anaerobic bacteria, small bowel bacterial overgrowth, Clostridium difficile colitis and also Giardia, which is common amongst children with SAM. Small cohort studies of metronidazole usage suggest there may be benefits for nutritional recovery in malnourished children. However, metronidazole can cause nausea and anorexia, potentially impairing recovery from malnutrition and may also rarely cause liver and neurological toxicity.

This multi-centre clinical trial will assess the efficacy of two interventions, ceftriaxone and metronidazole, on mortality and nutritional recovery in sick, severely malnourished children in a 2x2 factorial design. There will also be an analysis of antimicrobial resistance and an economic analysis. To extend our understanding of metronidazole and ceftriaxone pharmacokinetics, additional pharmacokinetic data for the dosing schedule used in the trial will be collected from 120 participants in a sub-study. The trial will be conducted at Kilifi County Hospital, Coast General Hospital, Mbagathi Hospital in Kenya and Mbale Regional Referral Hospital in Uganda. The trial will assess antimicrobial resistance that is carried by children in their intestines and in invasive bacterial isolates. A further sub-study will examine the relative costs of care for SAM for health facilities and for families, including antimicrobial usage will also be assessed. Clear data on the benefits, risks and costs of these antimicrobials will influence policy on case management and antimicrobial stewardship in this vulnerable population.

ELIGIBILITY:
Inclusion:

* Age 2 months to 13 years inclusive
* Severe malnutrition defined as:
* kwashiorkor at any age or:
* for children between 2 to 5 months: MUAC <11cm or weight-for length Z score <-3
* for children between 6 to 59 months: MUAC <11.5cm or weight-for length Z score <-3
* for children between 5 to 13 years: MUAC <11.5cm or BMI-for-age Z score <-3
* Admitted to hospital and eligible for intravenous antibiotics according to WHO guidelines
* Planning to remain within the hospital catchment area and willing to come for specified visits during the 90 day follow up period
* Informed consent provided by the parents/guardian

Exclusion:

* Known allergy or contraindication to penicillin, gentamicin, ceftriaxone or metronidazole
* A specific and documented clinical indication for another class of antibiotic
* Previously enrolled in this study

Ages: 2 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days after enrolment.
  Mortality is measured using source documents from medical records, verbal autopsy, or death or burial certificates in the community.

SECONDARY OUTCOMES:
Mortality during the first 7 days | 7 days
  Mortality during the first 7 days
Mortality during the first 30 days | 7 days
  Mortality during the first 30 days
Index admission inpatient mortality | Through index hospital admission, an average of 7 days.
  Mortality during the index hospitalisation, measured using inpatient records.
Mortality after discharge from index admission. | 90 days after enrolment
  Mortality occurring after discharge from the index hospital admission is measured using inpatient medical records, verbal autopsy, or death or burial certificates in the community.
Grade 4 toxicity | Up to 7 days following enrolment
  Grade 4 toxicity events are measured according to the Division of AIDS Tables for Grading the Severity of Adverse Events using medical records.
Serious adverse events | 90 days after enrolment.
  Serious adverse events are measured using inpatient and outpatient medical records.
Tolerability - relevant side effects during the first 7 day | 7 days
  Vomiting, diarrhoea, NG tube in place and convulsions during the first 7 days
Causes of death. | 90 days after enrolment
  Causes of death, as determined by an endpoint review committee.
Re-admission to hospital. | From discharge from hospital to 90 days after enrolment
  Re-admission to hospital defined as at least one overnight stay in a hospital or health facility are measured using inpatient records.
Duration of hospitalisation. | 90 days after enrolment.
  Total duration of hospitalisation is measured in days using inpatient records at the start and end of each admission to hospital.
Duration of administration of antibiotics. | 90 days after enrolment.
  Duration of administration of intravenous antibiotics measured using inpatient records.
Change in nutritional status | 90 days after enrolment.
  Change in nutritional status is measured using mid-upper arm circumference, weight-for-length, weight-for-age and length-for-age compared to at enrollment.
Faecal carriage of bacteria expressing Extended Spectrum Lactamase (ESBL) | Through study completion an average of 90 days.
  Faecal carriage of bacteria expressing Extended Spectrum Lactamase (ESBL) is measured using microbial culture and sensitivity testing of rectal swabs.

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkely, FRCPCH, Principal Investigator — KEMRI/Wellcome Trust Research Programme & University of Oxford
Locations (8):
- Kenya (7):
  - Kemri Wellcome Trust Research Programme, Kilifi, Coast Province
  - Kilifi County Hospital, Kilifi, Coast
  - KEMRI WT Clinical Trials Facility, Kilifi
  - Kilifi County Hospital, Kilifi
  - Coast General Hospital - Study site, Mombasa
  - Mbagathi District Hospital, Nairobi
  - Mbagathi Hospital, Nairobi
- Mbale Regional Referral Hospital, Mbale, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be considered by applying to the Data Governance Committee at CGMR,C Kilifi who will manage the process and ensure that appropriate ethical approval is in place and consent has been obtained for uses outside those given in this protocol:DGC@kemri-wellcome.org. Explanation of this eventuality will be included in the participant information and consent form. We intend to share anonymised data with the CHAIN network cohort study (KEMRI/SERU/CGMR-C /054/3318, OxTREC 34-16) which consists of institutions doing studies in malnourished children in Africa and South Asia; to upload anonymised bacterial and resistance sequences on recognised international repositories; and share anonymised bacterial sequence data relating to bacterial resistance with groups working an antimicrobial resistance in Africa and elsewhere.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years after study end, no end date foreseen
Access Criteria: Managed access. Apply to the Data Governance Committee: dgc@kemri-wellcome.org

REFERENCES:
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Acquah SE, Quaye L, Sagoe K, Ziem JB, Bromberger PI, Amponsem AA. Susceptibility of bacterial etiological agents to commonly-used antimicrobial agents in children with sepsis at the Tamale Teaching Hospital. BMC Infect Dis. 2013 Feb 18;13:89. doi: 10.1186/1471-2334-13-89. PMID 23419199
- [Background] Talbert A, Thuo N, Karisa J, Chesaro C, Ohuma E, Ignas J, Berkley JA, Toromo C, Atkinson S, Maitland K. Diarrhoea complicating severe acute malnutrition in Kenyan children: a prospective descriptive study of risk factors and outcome. PLoS One. 2012;7(6):e38321. doi: 10.1371/journal.pone.0038321. Epub 2012 Jun 4. PMID 22675542
- [Background] Heikens GT, Bunn J, Amadi B, Manary M, Chhagan M, Berkley JA, Rollins N, Kelly P, Adamczick C, Maitland K, Tomkins A; Blantyre Working Group. Case management of HIV-infected severely malnourished children: challenges in the area of highest prevalence. Lancet. 2008 Apr 12;371(9620):1305-7. doi: 10.1016/S0140-6736(08)60565-6. No abstract available. PMID 18406865
- [Background] Chimhuya S, Kambarami RA, Mujuru H. The levels of malnutrition and risk factors for mortality at Harare Central Hospital-Zimbabwe: an observation study. Cent Afr J Med. 2007 May-Aug;53(5-8):30-4. doi: 10.4314/cajm.v53i5-8.62612. PMID 20355679
- [Background] Fergusson P, Tomkins A. HIV prevalence and mortality among children undergoing treatment for severe acute malnutrition in sub-Saharan Africa: a systematic review and meta-analysis. Trans R Soc Trop Med Hyg. 2009 Jun;103(6):541-8. doi: 10.1016/j.trstmh.2008.10.029. Epub 2008 Dec 5. PMID 19058824
- [Background] Moisi JC, Gatakaa H, Berkley JA, Maitland K, Mturi N, Newton CR, Njuguna P, Nokes J, Ojal J, Bauni E, Tsofa B, Peshu N, Marsh K, Williams TN, Scott JA. Excess child mortality after discharge from hospital in Kilifi, Kenya: a retrospective cohort analysis. Bull World Health Organ. 2011 Oct 1;89(10):725-32, 732A. doi: 10.2471/BLT.11.089235. Epub 2011 Jul 13. PMID 22084510
- [Background] Berkley JA, Lowe BS, Mwangi I, Williams T, Bauni E, Mwarumba S, Ngetsa C, Slack MP, Njenga S, Hart CA, Maitland K, English M, Marsh K, Scott JA. Bacteremia among children admitted to a rural hospital in Kenya. N Engl J Med. 2005 Jan 6;352(1):39-47. doi: 10.1056/NEJMoa040275. PMID 15635111
- [Background] Trehan I, Goldbach HS, LaGrone LN, Meuli GJ, Wang RJ, Maleta KM, Manary MJ. Antibiotics as part of the management of severe acute malnutrition. N Engl J Med. 2013 Jan 31;368(5):425-35. doi: 10.1056/NEJMoa1202851. PMID 23363496
- [Background] Babirekere-Iriso E, Musoke P, Kekitiinwa A. Bacteraemia in severely malnourished children in an HIV-endemic setting. Ann Trop Paediatr. 2006 Dec;26(4):319-28. doi: 10.1179/146532806X152845. PMID 17132297
- [Background] Blomberg B, Manji KP, Urassa WK, Tamim BS, Mwakagile DS, Jureen R, Msangi V, Tellevik MG, Holberg-Petersen M, Harthug S, Maselle SY, Langeland N. Antimicrobial resistance predicts death in Tanzanian children with bloodstream infections: a prospective cohort study. BMC Infect Dis. 2007 May 22;7:43. doi: 10.1186/1471-2334-7-43. PMID 17519011
- [Background] Aiken AM, Mturi N, Njuguna P, Mohammed S, Berkley JA, Mwangi I, Mwarumba S, Kitsao BS, Lowe BS, Morpeth SC, Hall AJ, Khandawalla I, Scott JAG; Kilifi Bacteraemia Surveillance Group. Risk and causes of paediatric hospital-acquired bacteraemia in Kilifi District Hospital, Kenya: a prospective cohort study. Lancet. 2011 Dec 10;378(9808):2021-2027. doi: 10.1016/S0140-6736(11)61622-X. Epub 2011 Nov 29. PMID 22133536
- [Background] Woerther PL, Angebault C, Jacquier H, Hugede HC, Janssens AC, Sayadi S, El Mniai A, Armand-Lefevre L, Ruppe E, Barbier F, Raskine L, Page AL, de Rekeneire N, Andremont A. Massive increase, spread, and exchange of extended spectrum beta-lactamase-encoding genes among intestinal Enterobacteriaceae in hospitalized children with severe acute malnutrition in Niger. Clin Infect Dis. 2011 Oct;53(7):677-85. doi: 10.1093/cid/cir522. PMID 21890771
- [Background] Paterson DL. "Collateral damage" from cephalosporin or quinolone antibiotic therapy. Clin Infect Dis. 2004 May 15;38 Suppl 4:S341-5. doi: 10.1086/382690. PMID 15127367
- [Background] Jones KD, Hunten-Kirsch B, Laving AM, Munyi CW, Ngari M, Mikusa J, Mulongo MM, Odera D, Nassir HS, Timbwa M, Owino M, Fegan G, Murch SH, Sullivan PB, Warner JO, Berkley JA. Mesalazine in the initial management of severely acutely malnourished children with environmental enteric dysfunction: a pilot randomized controlled trial. BMC Med. 2014 Aug 14;12:133. doi: 10.1186/s12916-014-0133-2. PMID 25189855
- [Background] Ignatius R, Gahutu JB, Klotz C, Steininger C, Shyirambere C, Lyng M, Musemakweri A, Aebischer T, Martus P, Harms G, Mockenhaupt FP. High prevalence of Giardia duodenalis Assemblage B infection and association with underweight in Rwandan children. PLoS Negl Trop Dis. 2012;6(6):e1677. doi: 10.1371/journal.pntd.0001677. Epub 2012 Jun 12. PMID 22720102
- [Background] Heikens GT, Schofield WN, Christie CD, Gernay J, Dawson S. The Kingston Project. III. The effects of high energy supplement and metronidazole on malnourished children rehabilitated in the community: morbidity and growth. Eur J Clin Nutr. 1993 Mar;47(3):174-91. PMID 8458315
- [Background] Dubray C, Ibrahim SA, Abdelmutalib M, Guerin PJ, Dantoine F, Belanger F, Legros D, Pinoges L, Brown V. Treatment of severe malnutrition with 2-day intramuscular ceftriaxone vs 5-day amoxicillin. Ann Trop Paediatr. 2008 Mar;28(1):13-22. doi: 10.1179/146532808X270635. PMID 18318945
- [Background] Berkley JA, Ngari M, Thitiri J, Mwalekwa L, Timbwa M, Hamid F, Ali R, Shangala J, Mturi N, Jones KD, Alphan H, Mutai B, Bandika V, Hemed T, Awuondo K, Morpeth S, Kariuki S, Fegan G. Daily co-trimoxazole prophylaxis to prevent mortality in children with complicated severe acute malnutrition: a multicentre, double-blind, randomised placebo-controlled trial. Lancet Glob Health. 2016 Jul;4(7):e464-73. doi: 10.1016/S2214-109X(16)30096-1. Epub 2016 Jun 2. PMID 27265353
- [Background] Haybittle JL. Repeated assessment of results in clinical trials of cancer treatment. Br J Radiol. 1971 Oct;44(526):793-7. doi: 10.1259/0007-1285-44-526-793. No abstract available. PMID 4940475
- [Background] Peto R, Pike MC, Armitage P, Breslow NE, Cox DR, Howard SV, Mantel N, McPherson K, Peto J, Smith PG. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. I. Introduction and design. Br J Cancer. 1976 Dec;34(6):585-612. doi: 10.1038/bjc.1976.220. PMID 795448
- [Background] Standing JF, Ongas MO, Ogwang C, Kagwanja N, Murunga S, Mwaringa S, Ali R, Mturi N, Timbwa M, Manyasi C, Mwalekwa L, Bandika VL, Ogutu B, Waichungo J, Kipper K, Berkley JA; FLACSAM-PK Study Group. Dosing of Ceftriaxone and Metronidazole for Children With Severe Acute Malnutrition. Clin Pharmacol Ther. 2018 Dec;104(6):1165-1174. doi: 10.1002/cpt.1078. Epub 2018 Apr 19. PMID 29574688
- [Background] Ongas M, Standing J, Ogutu B, Waichungo J, Berkley JA, Kipper K. Liquid chromatography-tandem mass spectrometry for the simultaneous quantitation of ceftriaxone, metronidazole and hydroxymetronidazole in plasma from seriously ill, severely malnourished children. Wellcome Open Res. 2017 Jun 19;2:43. doi: 10.12688/wellcomeopenres.11728.2. eCollection 2017. PMID 29479566
- [Background] Williams PCM, Berkley JA. Guidelines for the treatment of severe acute malnutrition: a systematic review of the evidence for antimicrobial therapy. Paediatr Int Child Health. 2018 Nov;38(sup1):S32-S49. doi: 10.1080/20469047.2017.1409453. PMID 29790840
- [Background] Williams PCM, Isaacs D, Berkley JA. Antimicrobial resistance among children in sub-Saharan Africa. Lancet Infect Dis. 2018 Feb;18(2):e33-e44. doi: 10.1016/S1473-3099(17)30467-X. Epub 2017 Oct 9. PMID 29033034
- See also: Pocket book of hospital care for children Guidelines for the management of common illnesses with limited resources Author: World Health Organization — http://apps.who.int/iris/bitstream/10665/43206/1/9241546700.pdf